CLINICAL TRIAL: NCT02866799
Title: Effectiveness of an Intervention for Improving Drug Prescription in Primary Care Patients With Multimorbidity and Polypharmacy: Study Protocol of a Cluster Randomized Clinical Trial (Multi-PAP Project)
Brief Title: Multi-PAP: Improving Prescription in Primary Care Patients With Multimorbidity and Polypharmacy
Acronym: Multi-PAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Collaborators: Gerencia de Atención Primaria, Madrid (Other Government); Aragon Institute for Health Research (IIS Aragón) (Unknown); Andaluz Health Service (Other Government); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Alexandra Prados Torres, Medical Doctor, PhD, Instituto Aragones de Ciencias de la Salud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PI: 15/00572,15/00276,15/00996
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Multimorbidity; Polypharmacy; Other Diagnoses, Comorbidities, and Complications
Keywords: Multimorbidity; Primary Health Care; Polypharmacy; Comorbidity; Medication Adherence; Medication Appropriateness Index; Patient-Centered Care
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-PAP intervention (Experimental): Complex intervention with general practitioners and patients
  Interventions: Other: Multi-PAP; Other: Usual care
- Usual care (Active Comparator): Patients will receive the usual clinical care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Multi-PAP — Complex intervention based on the ARIADNE principles with two main components: 1) Training of general practitioners and 2) Patient centered clinical interview.
  Arms: Multi-PAP intervention
Other: Usual care — Patients will receive the usual clinical care based on current clinical practice guidelines.

SUMMARY:
This study assesses the effectiveness of a complex intervention in young-old patients with multimorbidity and polypharmacy aimed at improving physician drug prescription in primary care, measured by means of the Medication Appropriateness Index (MAI)-score at six 6 (T1) and 12 (T2) months from baseline compared to usual care.

DETAILED DESCRIPTION:
Design: Pragmatic cluster randomized clinical trial with 12 months follow-up.

Unit of randomization: general practitioner.

Unit of analysis: patient.

Setting: Primary Health Care Centres in three different Spanish Autonomous Communities (Aragón, Madrid and Andalucía).

Population: Patients 65-74 years of age with multimorbidity (3 or more chronic diseases) and polypharmacy (5 or more drugs taken for at least three months). N=400 patients (200 in each arm, 5 patients per physician) will be recruited by general practitioners before randomization.

Intervention: complex intervention.

Control group: usual care.

Variables: MAI, health care utilization, quality of life (Euroqol 5 Dimensions (5D-5L), drug therapy and adherence (Morisky-Green, Haynes-Sackett), clinical and socio-demographic factors. Economic appraisal variables: time spent training FPs, cost of teaching staff, time spent on physician-patient interviews, utilities measured using the EuroQol 5D-5L.

Analysis: All analyses will be carried out adhering to the intention-to-treat principle. Description of baseline characteristics. Basal comparison between groups. Analysis of main and secondary effectiveness (between-group difference in T1-T0 MAI score, with corresponding 95% Confidence Interval); multilevel analysis will be used to adjust models. Estimated quality-adjusted life years (QALYs) gained at the population level. Calculation of cost-utility ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65-74 years of age with multimorbidity (3 or more chronic diseases) and polypharmacy (5 or more drugs taken for at least three months).
* Informed consent.

Exclusion Criteria:

* Institutionalized patient at nursing homes or similar
* Life expectancy < 12 months

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 593 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Medication Appropriateness Index (MAI) score | Change from baseline MAI score at 6 months

SECONDARY OUTCOMES:
Medication Appropriateness Index (MAI) score | Change from baseline MAI score at 12 months
  Quality of Life
Morisky-Green questionnaire | Baseline, at six 6 months and at 12 months
  Therapeutic adherence questionnaire
Haynes-Sackett test | Baseline, at six 6 months and at 12 months
  Therapeutic adherence test
Euroqol 5D-5L questionnaire | Baseline, at six 6 months and at 12 months
Use of health services | at six 6 months and at 12 months
  Unscheduled and/or avoidable hospitalizations, use of emergency services and primary care (FP and nurse).
Medication safety | at six 6 months and at 12 months
  measured as the incidence of adverse drug reactions and potentially hazardous interactions, classified using the taxonomy proposed by Otero-López
Patient perception of shared decision-making | Baseline and at six 6 months and at 12 months
  measured using a single, multiple choice question, formulated ad hoc.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Prados-Torres, MD, PhD, Principal Investigator — Instituto Aragonés de Ciencias de la Salud (IACS); Daniel Prados-Torres, MD, PhD, Principal Investigator — Servicio Andaluz de Salud (Andaluz Health Service); Isabel Del Cura-González, MD, PhD, Principal Investigator — Gerencia de Atención Primaria, Madrid
Locations (3):
- Spain (3):
  - Málaga, Andalusia
  - Zaragoza, Aragon
  - Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prados-Torres A, Del Cura-Gonzalez I, Prados-Torres D, Lopez-Rodriguez JA, Leiva-Fernandez F, Calderon-Larranaga A, Lopez-Verde F, Gimeno-Feliu LA, Escortell-Mayor E, Pico-Soler V, Sanz-Cuesta T, Bujalance-Zafra MJ, Morey-Montalvo M, Boxo-Cifuentes JR, Poblador-Plou B, Fernandez-Arquero JM, Gonzalez-Rubio F, Ramiro-Gonzalez MD, Coscollar-Santaliestra C, Martin-Fernandez J, Barnestein-Fonseca MP, Valderas-Martinez JM, Marengoni A, Muth C; Multi-PAP Group. Effectiveness of an intervention for improving drug prescription in primary care patients with multimorbidity and polypharmacy: study protocol of a cluster randomized clinical trial (Multi-PAP project). Implement Sci. 2017 Apr 27;12(1):54. doi: 10.1186/s13012-017-0584-x. PMID 28449721
- [Background] Prados-Torres A, Del Cura-Gonzalez I, Prados-Torres JD, Leiva-Fernandez F, Lopez-Rodriguez JA, Calderon-Larranaga A, Muth C. [Multimorbidity in general practice and the Ariadne principles. A person-centred approach]. Aten Primaria. 2017 May;49(5):300-307. doi: 10.1016/j.aprim.2016.11.013. Epub 2017 Apr 17. Spanish. PMID 28427915
- [Background] Prados-Torres D, Del Cura-Gonzalez I, Prados-Torres A. [Towards a multimorbidity care model in Primary Care]. Aten Primaria. 2017 May;49(5):261-262. doi: 10.1016/j.aprim.2016.11.004. Epub 2017 Jan 11. No abstract available. Spanish. PMID 28089227
- [Result] Rogero-Blanco E, Lopez-Rodriguez JA, Sanz-Cuesta T, Aza-Pascual-Salcedo M, Bujalance-Zafra MJ, Cura-Gonzalez I; MultiPAP Group. Use of an Electronic Clinical Decision Support System in Primary Care to Assess Inappropriate Polypharmacy in Young Seniors With Multimorbidity: Observational, Descriptive, Cross-Sectional Study. JMIR Med Inform. 2020 Mar 3;8(3):e14130. doi: 10.2196/14130. Erratum In: JMIR Med Inform. 2020 Nov 19;8(11):e25678. doi: 10.2196/25678. PMID 32149715
- [Result] Prados-Torres A, Cura-Gonzalez ID, Prados-Torres JD, Muth C, Leiva-Fernandez F, Lopez-Rodriguez JA, Gonzalez-Rubio F. MULTIPAP Study: Improving healthcare for patients with multimorbidity. Br J Gen Pract. 2020 Jun;70(suppl 1):bjgp20X711257. doi: 10.3399/bjgp20X711257. PMID 32554653
- [Result] Lozano-Hernandez CM, Lopez-Rodriguez JA, Leiva-Fernandez F, Calderon-Larranaga A, Barrio-Cortes J, Gimeno-Feliu LA, Poblador-Plou B, Cura-Gonzalez ID; MULTIPAP GROUP. Social support, social context and nonadherence to treatment in young senior patients with multimorbidity and polypharmacy followed-up in primary care. MULTIPAP Study. PLoS One. 2020 Jun 24;15(6):e0235148. doi: 10.1371/journal.pone.0235148. eCollection 2020. PMID 32579616
- [Derived] Del Cura-Gonzalez I, Lopez-Rodriguez JA, Leiva-Fernandez F, Gimeno-Miguel A, Poblador-Plou B, Lopez-Verde F, Lozano-Hernandez C, Pico-Soler V, Bujalance-Zafra MJ, Gimeno-Feliu LA, Aza-Pascual-Salcedo M, Rogero-Blanco M, Gonzalez-Rubio F, Garcia-de-Blas F, Polentinos-Castro E, Sanz-Cuesta T, Castillo-Jimena M, Alonso-Garcia M, Calderon-Larranaga A, Valderas JM, Marengoni A, Muth C, Prados-Torres JD, Prados-Torres A; Multi-Pap Group. How to Improve Healthcare for Patients with Multimorbidity and Polypharmacy in Primary Care: A Pragmatic Cluster-Randomized Clinical Trial of the MULTIPAP Intervention. J Pers Med. 2022 May 6;12(5):752. doi: 10.3390/jpm12050752. PMID 35629175
- [Derived] Leiva-Fernandez F, Prados-Torres JD, Prados-Torres A, Del-Cura-Gonzalez I, Castillo-Jimena M, Lopez-Rodriguez JA, Rogero-Blanco ME, Lozano-Hernandez CM, Lopez-Verde F, Bujalance-Zafra MJ, Pico-Soler MV, Gimeno-Feliu LA, Poblador-Plou B, Martinez-Canavate MT, Muth C; MULTIPAP Group. Training primary care professionals in multimorbidity management: Educational assessment of the eMULTIPAP course. Mech Ageing Dev. 2020 Dec;192:111354. doi: 10.1016/j.mad.2020.111354. Epub 2020 Sep 15. PMID 32946885